CLINICAL TRIAL: NCT01334424
Title: Oxidative Stress in Robot-assisted Laparoscopic Radical Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Chang Gung Memorial Hospital, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: CGMH-IRB-98-2998B; CMRPG390841 (Other Grant/Funding Number: Chang Gung Memorial Hospital)
Record Dates: First submitted 2011-02-27; First posted 2011-04-13 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Oxidative Stress
Keywords: Robot assisted laparoscopic radical prostatectomy; Hypoperfusion reperfusion injury,; Propofol; oxidative stress
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- no propofol (Placebo Comparator): induction anesthesia with midazolam 0.2 - 0.3 mg/kg
  Interventions: Drug: propofol
- propofol induction (Experimental): induction anesthesia with propofol 2 - 2.5 mg/kg
  Interventions: Drug: propofol
- propofol maintenance (Experimental): induction anesthesia with midazolam 0.2 - 0.3 mg/kg and maintain anesthesia with propofol 2 mg/kg.h (maintenance dose)
  Interventions: Drug: propofol
- propofol induction and maintenance (Experimental): induction anesthesia with propofol 2 - 2.5 mg/ kg and maintain anesthesia with propofol 2 mg/kg.h (maintenance dose)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — 2-2.5 mg/kg for induction plus or not plus 2 mg/kg.h for maintenance

SUMMARY:
Gut hypoperfusion - reperfusion injury is an unavoidable event at the end of laparoscopic surgery. It produces oxidative stress (reactive oxygen species). Malondialdehyde have been demonstrated to be a reliable biomarker for the evaluation of oxidative stress in vivo. Propofol (2, 6 - diisopropylphenol), a highly liposoluble anaesthetic, has a potent antioxidant activity against lipid peroxidation in both in vitron and in vivo studies. On the basis of this knowledge, the investigators hypothesized that propofol has preventive effect for gut hypoperfusion - reperfusion induced injury in robot-assisted laparoscopic radical prostatectomy.

DETAILED DESCRIPTION:
Increased intrabdominal pressure is associated with pneumoperitoneum for laparoscopic procedures and is one of the main factors in impairment of splanchnic perfusion by compressing vessels. An hypoperfusion - reperfusion human model is observed during and soon after laparoscopic surgery. After deflation of the abdomen, intrabdominal pressure and splanchnic blood flow normalize, representing reperfusion.

Reactive oxygen species is produced in metabolic and physiologic processes, and harmful oxidative reactions may occur in organisms that remove them via enzymatic and nonenzymatic antioxidative mechanisms.

Propofol (2, 6 - diisopropylphenol), a highly liposoluble anaesthetic, has a potent antioxidant activity against lipid peroxidation in both in vitron and in vivo studies. Propofol also attenuates ischemia - reperfusion induced lipid peroxidation in humans. On the basis of this knowledge, we hypothesized that propofol has preventive effect for gut hypoperfusion - reperfusion induced injury in robot-assisted laparoscopic radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving robot-assisted laparoscopic radical prostatectomy in ASA II-III physical status

Exclusion Criteria:

* history of sepsis or shock, clinically relevant cardiopulmonary disease, persistent tobacco abuse, recent antioxidant or vasoconstrictor use

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Amount of Malondialdehyde in plasma | one day

CONTACTS AND LOCATIONS:
Overall Officials: Chiao-Fen Luo, MD, Principal Investigator — Dept. of Anesthesiology, Chang Gung Memorial Hospital
Locations (1):
- Dept. of Anesthesiology, Chang Gung Memorial Hospital, Taoyuan District, Taiwan